CLINICAL TRIAL: NCT03600753
Title: Characterization of Respiratory Microbiota in Susceptibility to Viral Respiratory Infections Using Metagenomic and Culturomic Approach
Brief Title: Characterization of Respiratory Microbiota in Susceptibility to Viral Respiratory Infections
Acronym: RESPIBIOTE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2017-23
Record Dates: First submitted 2018-07-03; First posted 2018-07-26 (Actual); Last update posted 2018-07-26 (Actual); Status verified 2018-06

CONDITIONS: Viral Respiratory Infection
MeSH Terms: interventions — malacidins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- symptomatic patients (Experimental): symptomatic patients with viral respiratory infection harboring positive qPCR for respiratory virus (influenza A or B, RSV, rhinovirus, metapneumovirus) A pharyngeal and a nasal swabs will be performed for each patient. Culturomic and metagenomic analyses will be performed
  Interventions: Other: culturomic; Other: Metagenomic
- asymptomatic patients (Active Comparator): symptomatic patients with viral respiratory infection with positive qPCR for respiratory virus.
  A pharyngeal and a nasal swabs will be performed for each patient. Culturomic and metagenomic analyses will be performed
  Interventions: Other: culturomic; Other: Metagenomic
- healthy subjects (Other): Control group of healthy patients. A pharyngeal and a nasal swabs will be performed for each patient. Culturomic and metagenomic analyses will be performed
  Interventions: Other: culturomic; Other: Metagenomic

INTERVENTIONS:
Other: culturomic — Culturomic is a high-throughput culture strategy based on the multiplication of culture conditions coupled with the rapid identification of bacteria by MALDI-TOF (Matrix-Assisted Laser Desorption / Ionization-Time-Of-Flight) mass spectrometry
Other: Metagenomic — Metagenomics is an high throughput sequencing and will be performed using Miseq ( Illumina technology) targeting the V3-V4 hypervariable regions of the 16S RNA gene.

SUMMARY:
The role of the nasopharyngeal mucosal microbiota has recently been emphasized in respiratory diseases. The hypothesis that respiratory infections are linked to an imbalance of the nasopharyngeal microbiota has recently emerged and some studies show a link between the respiratory microbiota, the susceptibility to viral respiratory infections and the severity induced. In a preliminary work on the respiratory microbiota from 225 patients and 48 controls, the investigators found a decrease in the richness and biodiversity of the nasopharyngeal microbiota in patients with a respiratory viral infection as well as an enrichment of their respiratory flora in pathogenic bacteria.

Interestingly, these recent years, the development of qPCR for virus diagnosis showed a substantial proportion of asymptomatic carriers of viruses suggesting that the nasopharyngeal microbiota may play a critical role in the genesis and clinical expression of viral respiratory infection, challenging Koch's postulate.

The principal objectives of this study are to compare the respiratory microbiota between symptomatic patients with respiratory viral infection and asymptomatic carrier of virus. The aim is to determine the existence of respiratory microbiota profiles associated with the occurrence of viral respiratory infections influencing the clinical expression of virus and to determine the role of the respiratory microbiota in the occurrence of bacterial superinfection which will justify an early antibiotic treatment.

The investigators will include 35 symptomatic patients with viral respiratory infection harboring positive qPCR for respiratory virus (influenza A or B, RSV, rhinovirus, metapneumovirus), 35 asymptomatic patients with positive qPCR for respiratory virus and 30 healthy subjects (controls). A pharyngeal and a nasal swabs will be performed for each patient. All the samples will be analyse by culturomics and metagenomic. Culturomic is a high-throughput culture strategy based on the multiplication of culture conditions coupled with the rapid identification of bacteria by MALDI-TOF (Matrix-Assisted Laser Desorption / Ionization-Time-Of-Flight) mass spectrometry.Metagenomics is an high throughput sequencing and will be performed using Miseq ( Illumina technology) targeting the V3-V4 hypervariable regions of the 16S RNA gene.

DETAILED DESCRIPTION:
The role of the nasopharyngeal mucosal microbiota has recently been emphasized in respiratory diseases. The hypothesis that respiratory infections are linked to an imbalance of the nasopharyngeal microbiota has recently emerged and some studies show a link between the respiratory microbiota, the susceptibility to viral respiratory infections and the severity induced. In a preliminary work on the respiratory microbiota from 225 patients and 48 controls, the investigators found a decrease in the richness and biodiversity of the nasopharyngeal microbiota in patients with a respiratory viral infection as well as an enrichment of their respiratory flora in pathogenic bacteria.

Interestingly, these recent years, the development of qPCR for virus diagnosis showed a substantial proportion of asymptomatic carriers of viruses suggesting that the nasopharyngeal microbiota may play a critical role in the genesis and clinical expression of viral respiratory infection, challenging Koch's postulate.

The principal objectives of this study are to compare the respiratory microbiota between symptomatic patients with respiratory viral infection and asymptomatic carrier of virus. The aim is to determine the existence of respiratory microbiota profiles associated with the occurrence of viral respiratory infections influencing the clinical expression of virus and to determine the role of the respiratory microbiota in the occurrence of bacterial superinfection which will justify an early antibiotic treatment.

The investigators will include 35 symptomatic patients with viral respiratory infection harboring positive qPCR for respiratory virus (influenza A or B, RSV, rhinovirus, metapneumovirus), 35 asymptomatic patients with positive qPCR for respiratory virus and 30 healthy subjects (controls). A pharyngeal and a nasal swabs will be performed for each patient. All the samples will be analyse by culturomics and metagenomic. Culturomic is a high-throughput culture strategy based on the multiplication of culture conditions coupled with the rapid identification of bacteria by MALDI-TOF (Matrix-Assisted Laser Desorption / Ionization-Time-Of-Flight) mass spectrometry.Metagenomics is an high throughput sequencing and will be performed using Miseq ( Illumina technology) targeting the V3-V4 hypervariable regions of the 16S RNA gene.

The precise characterization of the respiratory microbiota in patients with viral respiratory infections is still incomplete. Our work is original because it will combine innovative and complementary techniques of culturomics and metagenomics for the exhaustive study of the respiratory microbiota associated with respiratory viral disease.

ELIGIBILITY:
Inclusion Criteria:

* Adult > 18 years
* Hospitalized patients with respiratory viral infection diagnosed by qPCR and / or rapid tests
* Contact cases (parent, sister, brother, ...) of patients presenting with viral respiratory infection
* No one has expressed opposition to the processing of personal data
* Person who had been informed and had not expressed his opposition to participate in the study

Exclusion Criteria:

* Minor patient
* Subject who take antibiotic in the 3 weeks before the viral respiratory infection
* Presence of another non-respiratory bacterial infection
* Vulnerable person: Minor, person under guardianship, or deprived of liberty by a judicial or administrative decision

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-09-01 (Estimated); Primary Completion 2021-02 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
standard microbiological diagnosis of virology | 30 months
  qPCR influenza A, influenza B, rhinovirus, metapneumovirus and respiratory syncythial virus will be performed according to the laboratory protocol by PCR or immunochromatographic test.
Bacterial metagenomics | 30 months
  The composition of the respiratory microbiota will be established by high-throughput sequencing of the V3-V4 hypervariable regions of the 16S rRNA gene by Miseq (Illumina)
culturomic | 30 months
  Culturomic is a high-throughput culture strategy based on the multiplication of culture conditions coupled with the rapid identification of bacteria by MALDI-TOF (Matrix-Assisted Laser Desorption / Ionization-Time-Of-Flight) mass spectrometry ( 14). In the event of an insufficient identification score by MALDI-TOF, the strains are identified by molecular techniques, in particular by sequencing of the 16S rRNA.

SECONDARY OUTCOMES:
bacteria present in the respiratory flora in healthy group | 30 months
  Name of bacteria present in the resoiratory flora in healthy group
bacteria present in the respiratory flora of patients | 30 months
  Name of bacteria in the respiratory flora of patients with viral respiratory infection Identification mill be performed using culture approach.
Prognostic factors of viral respiratory infections | 30 months
  Prognostic factors (risk factors or protective factors) of viral respiratory infections by the identification of bacteria that play a protective or deleterious role in the occurrence of viral respiratory infection.

CONTACTS AND LOCATIONS:
Overall Officials: EMILIE GARRIDO PRADALIE, Study Director — APHM
Locations (1):
- Assistance Publique Des Hopitaux de Marseille, Marseille, PACA, France